CLINICAL TRIAL: NCT07371221
Title: Ultrasound-Guided Nerve Hydrodissection With 5% Dextrose in Carpal Tunnel Syndrome: A Prospective Study
Brief Title: Ultrasound-Guided Dextrose Hydrodissection of the Median Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nafiz Korez Sincan State Hospital (Other Government)
Responsible Party: Principal Investigator, Sevgi Esra Ozdemir Tekes, Medical Doctor, Dr. Nafiz Korez Sincan State Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-09
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel syndrome; hydrodissection; Microvascular imaging; ultrasound guided injection; median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective, non-randomized interventional study. All participants receive ultrasound-guided median nerve hydrodissection with 5% dextrose, and outcomes are measured before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-Guided Dextrose Median Nerve Hydrodissection (Experimental): Participants in this arm undergo a single session of ultrasound-guided median nerve hydrodissection using 5% dextrose solution. The procedure is performed under aseptic conditions with real-time ultrasound guidance to visualize the median nerve and surrounding anatomical structures within the carpal tunnel. The injectate is administered to mechanically separate the median nerve from adjacent tissues.
  Interventions: Procedure: Ultrasound-Guided Median Nerve Hydrodissection with 5% Dextrose

INTERVENTIONS:
Procedure: Ultrasound-Guided Median Nerve Hydrodissection with 5% Dextrose — This intervention consists of a single-session ultrasound-guided hydrodissection of the median nerve using 5% dextrose solution in patients with mild and moderate carpal tunnel syndrome. The procedure is performed under aseptic conditions by trained physicians using a high-frequency linear ultrasound transducer. Real-time in-plane imaging is used to visualize the median nerve and surrounding structures, and the injectate is administered via an ulnar approach to mechanically separate the median nerve from adjacent connective tissues within the carpal tunnel. Participants are monitored for any procedure-related adverse events during and after the intervention.

SUMMARY:
The goal of this clinical trial is to evaluate the clinical and ultrasonographic outcomes of ultrasound-guided median nerve hydrodissection with 5% dextrose in patients with mild and moderate carpal tunnel syndrome.

The main questions it aims to answer are:

* Does ultrasound-guided dextrose hydrodissection improve pain and functional status in patients with carpal tunnel syndrome?
* Does this procedure lead to changes in ultrasonographic parameters of the median nerve?
* Is ultrasound-guided dextrose hydrodissection a safe procedure in this patient population?

Participants will:

* Undergo a single session of ultrasound-guided median nerve hydrodissection with 5% dextrose
* Be evaluated before the procedure and at 1-month and 3-month follow-up visits using clinical outcome measures and ultrasound assessment
* Be monitored for any procedure-related adverse events

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy of the upper extremity and is caused by compression of the median nerve within the carpal tunnel. Conservative treatment options are commonly preferred in patients with mild to moderate CTS. Ultrasound-guided interventions have gained increasing attention due to their ability to provide real-time visualization of anatomical structures and improve procedural accuracy and safety.

Ultrasound-guided median nerve hydrodissection is a minimally invasive technique that aims to mechanically separate the median nerve from surrounding tissues within the carpal tunnel, potentially reducing nerve compression and improving nerve mobility. The use of 5% dextrose solution has been suggested to provide both mechanical and potential neuromodulatory effects, which may contribute to symptom relief.

In this prospective study, patients diagnosed with mild and moderate CTS undergo ultrasound-guided median nerve hydrodissection using 5% dextrose. All procedures are performed under aseptic conditions by experienced physicians trained in ultrasound-guided interventions. A high-frequency linear ultrasound transducer is used to visualize the median nerve and surrounding anatomical structures at the level of the carpal tunnel. Hydrodissection is performed using an in-plane technique, which allows for continuous visualization of the needle and injectate during the procedure.

Participants receive a single-session ultrasound-guided hydrodissection, during which the injectate is administered to separate the median nerve from adjacent connective tissues. The procedure is conducted according to a standardized protocol to ensure consistency across all participants.

Clinical and ultrasonographic assessments are performed at baseline, and at 1-month and 3-month follow-up visits after the ultrasound-guided injection. Patients are monitored for any procedure-related adverse events throughout the study period. The study aims to evaluate changes in clinical symptoms and ultrasound findings following the intervention, as well as to assess the safety profile of ultrasound-guided dextrose hydrodissection in patients with mild and moderate CTS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Electrophysiologically confirmed mild to moderate CTS on electroneuromyography (ENMG)
* Paresthesia or dysesthesia that worsens at night or with repetitive wrist movement
* Presence of at least one of the following clinical findings:

  1. Numbness in the median nerve distribution
  2. Decreased hand strength or thenar muscle weakness
  3. Positive Phalen's test and/or Tinel's sign
* Pain intensity of ≥3 on the Visual Analog Scale (VAS)

Exclusion Criteria:

* Previous carpal tunnel surgery
* Severe CTS on ENMG
* Polyneuropathy
* Pregnancy
* Injections in the same area within the last 3 months
* Peripheral nerve injury, thoracic outlet syndrome, cervical radiculopathy, brachial plexopathy
* Traumatic hand injury in the last 2 years
* Inflammatory rheumatological disease
* Thyroid and autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Baseline, 1 month and 3 months
  The severity of pain in the fingers over the past week was measured using a 10-cm Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in Vascularity Index of the Median Nerve | Baseline, 1 month and 3 months
  The Vascularity Index (VI) is a quantitative ultrasonographic measure of intraneural microvascularity of the median nerve. The VI is calculated as a percentage value ranging from 0 to 100, representing the proportion of pixels containing vascular signals within a predefined rectangular region of interest (ROI). Higher VI values indicate increased intraneural microvascularity and represent a worse disease-related finding.
Change in median nerve cross-sectional area | Baseline, 1 month and 3 months
  The cross-sectional area (CSA) of the median nerve was evaluated using ultrasonography by measuring the nerve at the thickest visible level within the carpal tunnel.
Change in Boston Carpal Tunnel Questionnaire | Baseline, 1 month and 3 months
  The Boston Carpal Tunnel Questionnaire (BCTQ) consists of two subscales: the Symptom Severity Scale (11 items), which assesses the intensity of CTS-related symptoms, and the Functional Status Scale (8 items), which evaluates the degree of difficulty in performing daily activities. Each item is scored on a 5-point scale ranging from 1 to 5, with higher scores indicating greater symptom severity in the Symptom Severity Scale and greater functional impairment in the Functional Status Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Suheyla Dal Erdogan, Medical Doctor, Study Chair — Dr. Nafiz Korez Sincan State Hospital; Sevgi Esra Ozdemir Tekes, Principal Investigator — Dr. Nafiz Korez Sincan State Hospital
Locations (1):
- Dr. Nafiz Korez Sincan State Hospital, Ankara, Ankara, Turkey (Türkiye)